CLINICAL TRIAL: NCT04760847
Title: Intermittent Fasting as a Primary Means for Improving Quality of Life for Acute and Chronic Pancreatitis
Brief Title: Intermittent Fasting for Pancreatitis
Acronym: IFPanc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20201373
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pancreatitis; Pancreatitis, Acute; Pancreatitis, Chronic; Pancreas Disease; Acute Recurrent Pancreatitis
Keywords: pancreatitis; acute pancreatitis; acute recurrent pancreatitis; chronic pancreatitis; fasting; intermittent fasting
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic; Pancreatic Diseases; Fasting; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The control group will have 32 patients and the group undergoing IF will have 32 patients (for both recurrent acute and chronic pancreatitis); the randomization is 1:1; IF versus control. Sixty four subjects will be enrolled at UH for a total of 64 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting (Experimental): Patients in Group A will then receive information regarding intermittent fasting, which would include fasting for a 16-hour period each day, followed by ingestion of an appropriate number of calories for the remaining part of the day.
  Interventions: Other: Intermittent Fasting
- Control (Active Comparator): These subjects will undergo standard caloric dietary guidance. Patients in group B will also be given the above information, though not be asked to intermittently fast.
  Interventions: Other: No intermittent fasting

INTERVENTIONS:
Other: Intermittent Fasting — These subjects will will then receive information regarding intermittent fasting, which would include fasting for a 16-hour period each day, followed by ingestion of an appropriate number of calories for the remaining part of the day. See attached IF Quick Facts for details provided to the patient.
  Arms: Intermittent Fasting
Other: No intermittent fasting — These subjects will undergo standard caloric dietary guidance. Patients in group B will also be given the above information, though not be asked to intermittently fast
  Arms: Control

SUMMARY:
The purpose of this research is to compare intermittent fasting with a standard diet approach for improving the quality of life related to your pancreas disease. Our hope is to improve your symptoms and prevent you from needing to go into the hospital for pancreas-related issues.

DETAILED DESCRIPTION:
Fasting is a classic means for religious discipline, yet recently regaining favor in the medical landscape. Numerous studies have come forth, both in animals and humans outlining the benefit of intermittent fasting (IF) on various disease states and longevity. Though a relatively complex cellular process, fasting for at least 8-12 hours has been shown to lead to fatty acid release from a patient's adipose storage. These fatty acids then shuttle to the liver, where they are converted to ketones such as beta-hydroxybutyrate and acetoacetate.

Ketones are then utilized for energy sources in the heart, brain and skeletal muscle tissue. The energy produced (ATP), then leads to increase in the cellular powerhouses, the mitochondria and autophagy or cell recycling. This cellular recycling is one main way in which IF has proven benefit for inflammatory conditions and in cancer care.

Furthermore, reductions in amino acids and glucose due to fasting and reliance on ketones as energy, lead to down regulation of the membrane target of rapamycin (mTOR) pathway. Much is known regarding the mTOR pathway. Down regulation of mTOR is associated with increased autophagy (as above), lower protein and lipid synthesis, ribosome and lysosome creation (cell shuttles) and lowered energy use.

Specific to the pancreas, mTOR down regulation has been shown to lower protein synthesis with the pancreas, caused by cholecystokinin (CCK), a pancreas stimulating hormone.2 The effect of this leads to lower pancreatic enzymes secretion. Inhibition of mTOR also lowers the generation of fibroblasts, the scar-tissue cells within the pancreas, leading to less scar-formation.3 Scar tissue formation is a vital part of morbidity and complications for patients with chronic pancreatitis.

Pancreatic disease-modulation has also been evaluated in regard to the mTOR pathway.4 For pancreatic cancer, rapamycin a mTOR inhibitor have been implicated as targets for chemotherapy. Clinical trials have shown benefit for pancreatic cancer cases given rapamycin in concert with other chemotherapeutic medications.5 For acute, chronic pancreatitis and post-ndoscopic retrograde cholangiopancreatopgraphy (ERCP) pancreatitis, mTOR is usually activated.6 In particular, blocking the mTOR pathway can favor autophagy, limit cell death (apoptosis) and hence necrosis of the pancreas. Necrosis in pancreatitis, leads to complex disease, possess a higher mortality, organ failure, and can make the clinical course more complicated. Therefore, the mTOR pathway has been implicated as a potential therapeutic target to ameliorate disease course and severity.4,7,8 The purpose of this study is to evaluate IF as a means for limiting disease severity with people who have recurrent acute pancreatitis and chronic pancreatitis. Our hypothesis is that IF will improve pancreatic-disease related quality of life.1

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Recurrent acute pancreatitis defined by greater than 2 episodes of pancreatitis, defined by:

abdominal pain and either amylase or lipase > 3 x the upper limit of normal, imaging suggestive of, separated by time

* Anatomy of chronic pancreatitis defined by Rosemont criterion9 or on imaging (CT, MRI)
* Pancreatic exocrine insufficiency defined by a pancreatic elastase < 200 ug/g stool10

Exclusion Criteria:

* Age < 18 years
* Pregnant Patients
* Age > 80 years
* Patients who cannot consent for themselves
* Glycogen storage disease
* Insulinoma or hypoglycemic state
* Active alcohol abuse
* Alcohol induced acute pancreatitis
* Gallstone induced acute pancreatitis
* Pancreatic solid neoplasm
* Patients with diabetes
* Patients on beta blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pancreas related Quality of Life Index (PANQALI) | 24 weeks
  Pancreas related Quality of Life Index (PANQALI) is pancreas related quality of life index scale from 0 (lowest or better disease activity) to 90 (highest or worse disease activity)

SECONDARY OUTCOMES:
Pain scores | 24 weeks
  standard score from 0-10 (0 no pain, 10 worst pain)
Oral Morphine Equivalent Daily Dosing | 24 weeks
  total dose of opiates taken converted into morphine in milligrams
Patient weight | 24 weeks
  pounds
Patient Body mass index | 24 weeks
  pounds/inch squared
Vitamin D 25-OH levels | 24 weeks
  levels of vitamin D 25-OH in nanograms/milliLiter
stool pancreatic elastase levels | 24 weeks
  stool elastase level in micrograms/gram
Readmissions | 24 weeks
  number of participants that need to seek medical care
Length of Stay | 24 weeks
  days requiring medical care

CONTACTS AND LOCATIONS:
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wassef W, DeWitt J, McGreevy K, Wilcox M, Whitcomb D, Yadav D, Amann S, Mishra G, Alkaade S, Romagnuolo J, Stevens T, Vargo J, Gardner T, Singh V, Park W, Hartigan C, Barton B, Bova C. Pancreatitis Quality of Life Instrument: A Psychometric Evaluation. Am J Gastroenterol. 2016 Aug;111(8):1177-86. doi: 10.1038/ajg.2016.225. Epub 2016 Jun 14. PMID 27296943
- [Background] Crozier SJ, Sans MD, Guo L, D'Alecy LG, Williams JA. Activation of the mTOR signalling pathway is required for pancreatic growth in protease-inhibitor-fed mice. J Physiol. 2006 Jun 15;573(Pt 3):775-86. doi: 10.1113/jphysiol.2006.106914. Epub 2006 Apr 13. PMID 16613881
- [Background] Yang J, Waldron RT, Su HY, Moro A, Chang HH, Eibl G, Ferreri K, Kandeel FR, Lugea A, Li L, Pandol SJ. Insulin promotes proliferation and fibrosing responses in activated pancreatic stellate cells. Am J Physiol Gastrointest Liver Physiol. 2016 Oct 1;311(4):G675-G687. doi: 10.1152/ajpgi.00251.2016. Epub 2016 Sep 8. PMID 27609771
- [Background] Bellizzi AM, Bloomston M, Zhou XP, Iwenofu OH, Frankel WL. The mTOR pathway is frequently activated in pancreatic ductal adenocarcinoma and chronic pancreatitis. Appl Immunohistochem Mol Morphol. 2010 Oct;18(5):442-7. doi: 10.1097/PAI.0b013e3181de115b. PMID 20661135
- [Background] Javle MM, Shroff RT, Xiong H, Varadhachary GA, Fogelman D, Reddy SA, Davis D, Zhang Y, Wolff RA, Abbruzzese JL. Inhibition of the mammalian target of rapamycin (mTOR) in advanced pancreatic cancer: results of two phase II studies. BMC Cancer. 2010 Jul 14;10:368. doi: 10.1186/1471-2407-10-368. PMID 20630061
- [Background] Law R, Leal C, Dayyeh BA, Leise MD, Balderramo D, Baron TH, Cardenas A. Role of immunosuppression in post-endoscopic retrograde cholangiopancreatography pancreatitis after liver transplantation: a retrospective analysis. Liver Transpl. 2013 Dec;19(12):1354-60. doi: 10.1002/lt.23758. PMID 24115362
- [Background] Ji L, Li L, Qu F, Zhang G, Wang Y, Bai X, Pan S, Xue D, Wang G, Sun B. Hydrogen sulphide exacerbates acute pancreatitis by over-activating autophagy via AMPK/mTOR pathway. J Cell Mol Med. 2016 Dec;20(12):2349-2361. doi: 10.1111/jcmm.12928. Epub 2016 Jul 15. PMID 27419805
- [Background] Wu XM, Ji KQ, Wang HY, Zhao Y, Jia J, Gao XP, Zang B. MicroRNA-339-3p alleviates inflammation and edema and suppresses pulmonary microvascular endothelial cell apoptosis in mice with severe acute pancreatitis-associated acute lung injury by regulating Anxa3 via the Akt/mTOR signaling pathway. J Cell Biochem. 2018 Aug;119(8):6704-6714. doi: 10.1002/jcb.26859. Epub 2018 Apr 25. PMID 29693276 (Retraction: PMID 34289164 J Cell Biochem. 2021 Nov;122 Suppl 1:S107)
- [Background] Conwell DL, Lee LS, Yadav D, Longnecker DS, Miller FH, Mortele KJ, Levy MJ, Kwon R, Lieb JG, Stevens T, Toskes PP, Gardner TB, Gelrud A, Wu BU, Forsmark CE, Vege SS. American Pancreatic Association Practice Guidelines in Chronic Pancreatitis: evidence-based report on diagnostic guidelines. Pancreas. 2014 Nov;43(8):1143-62. doi: 10.1097/MPA.0000000000000237. PMID 25333398
- [Background] Herzig KH, Purhonen AK, Rasanen KM, Idziak J, Juvonen P, Phillps R, Walkowiak J. Fecal pancreatic elastase-1 levels in older individuals without known gastrointestinal diseases or diabetes mellitus. BMC Geriatr. 2011 Jan 25;11:4. doi: 10.1186/1471-2318-11-4. PMID 21266058
- [Background] Han S, Patel B, Min M, Bocelli L, Kheder J, Wachholtz A, Wassef W. Quality of life comparison between smokers and non-smokers with chronic pancreatitis. Pancreatology. 2018 Apr;18(3):269-274. doi: 10.1016/j.pan.2018.02.012. Epub 2018 Feb 26. PMID 29500114
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Corley BT, Carroll RW, Hall RM, Weatherall M, Parry-Strong A, Krebs JD. Intermittent fasting in Type 2 diabetes mellitus and the risk of hypoglycaemia: a randomized controlled trial. Diabet Med. 2018 May;35(5):588-594. doi: 10.1111/dme.13595. Epub 2018 Feb 27. PMID 29405359